CLINICAL TRIAL: NCT06292052
Title: Relation Between Tumor-draining Lymph Nodes Metastasis Pattern and Non-small Cell Lung Cancer Neoadjuvant Immunotherapy Effectiveness: A Retrospective Multi-institutional Cohort Analysis
Brief Title: Relation Between Tumor-draining Lymph Nodes Metastasis Pattern and Non-small Cell Lung Cancer Neoadjuvant Immunotherapy Effectiveness
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Collaborators: Jiangmen Central Hospital (Other); Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Hao Long, Professor, Sun Yat-sen University
Other Study IDs: NSCLC-TDLN-001
Record Dates: First submitted 2024-02-23; First posted 2024-03-04 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Immunotherapy; Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Neoadjuvant immunochemotherapy NSCLC group: NSCLC patients who received neoadjuvant immunochemotherapy and underwent surgery.
  Interventions: Drug: Immunotherapy

INTERVENTIONS:
Drug: Immunotherapy — Received neoadjuvant chemotherapy plus immunotherapy
  Other Names: Chemotherapy

SUMMARY:
The goal of this retrospective cohort analysis is to discover the impact of the involvement extent of tumor-draining lymph nodes (TDLNs) in patients who received neoadjuvant immunochemotherapy. The main question it aims to answer is the role of TDLN in the prediction of treatment effectiveness. Researches will compare tumor-draining lymph nodes metastasis (mTDLNs) group and non-draining lymph nodes metastasis (mNDLNs) group to see whether different metastatic patterns of mediastinal lymph nodes can indicate the treatment effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* pathologically-confirmed diagnosis of NSCLC by pretreatment biopsy
* clinically staged as T1-4N0-2M0
* having undergo neoadjuvant chemoimmunotherapy
* the agents of immune checkpoint inhibitors (ICIs) belong to PD-1/L1 inhibitors
* having undergo surgery with lymph nodes (LNs) dissection
* having postoperative pathology reports with evaluation of primary tumor and LNs response
* having accessible pretreatment and preoperative radiology examinations imaging or reports

Exclusion Criteria:

* using PD-1/L1 inhibitors in the phase of clinical trials
* the agents of neoadjuvant therapy including angiogenesis inhibitors
* having undergone radiotherapy to treat primary tumor or metastatic LNs before surgery

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with resectable NSCLC (clinically staged as T1-4N0-2M0) who underwent neoadjuvant chemoimmunotherapy followed by surgery between January 2017 and January 2024 in Sun Yat-sen University Cancer Center were retrospectively reviewed.
Sampling Method: Non-Probability Sample
Enrollment: 209 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Complete pathologic response | through study completion, an average of 3 months
  Tumors with 0% viable tumor cells

SECONDARY OUTCOMES:
Major pathologic response | through study completion, an average of 3 months
  Tumors with ≤10% viable tumor cells
Complete pathologic response in lymph nodes | through study completion, an average of 3 months
  Tumors with 0% viable tumor cells in lymph nodes

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
The data will upload to ResMan after publication.

REFERENCES:
- [Result] Rahim MK, Okholm TLH, Jones KB, McCarthy EE, Liu CC, Yee JL, Tamaki SJ, Marquez DM, Tenvooren I, Wai K, Cheung A, Davidson BR, Johri V, Samad B, O'Gorman WE, Krummel MF, van Zante A, Combes AJ, Angelo M, Fong L, Algazi AP, Ha P, Spitzer MH. Dynamic CD8+ T cell responses to cancer immunotherapy in human regional lymph nodes are disrupted in metastatic lymph nodes. Cell. 2023 Mar 16;186(6):1127-1143.e18. doi: 10.1016/j.cell.2023.02.021. PMID 36931243
- [Result] Prokhnevska N, Cardenas MA, Valanparambil RM, Sobierajska E, Barwick BG, Jansen C, Reyes Moon A, Gregorova P, delBalzo L, Greenwald R, Bilen MA, Alemozaffar M, Joshi S, Cimmino C, Larsen C, Master V, Sanda M, Kissick H. CD8+ T cell activation in cancer comprises an initial activation phase in lymph nodes followed by effector differentiation within the tumor. Immunity. 2023 Jan 10;56(1):107-124.e5. doi: 10.1016/j.immuni.2022.12.002. Epub 2022 Dec 28. PMID 36580918